CLINICAL TRIAL: NCT06140953
Title: Evaluation of Potential Benefits of Trimetazidine in the Management of Patients With Metabolic Associated Steatotic Liver Disease (MASLD)
Brief Title: Benefits of Trimetazidine in MASLD Patients
Acronym: MASLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Maha youssif, principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-H-phBSU-23059
Record Dates: First submitted 2023-10-26; First posted 2023-11-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Associated Fatty Liver Disease
Keywords: trimetazidine in MASLD
MeSH Terms: interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (conventional treatment + placebo tablet) (Placebo Comparator): placebo tablet (inert substance) + Weight reduction and life style modification(modification in diet like decrease lipids intak).pateints will recieve their conventional therapy
  Interventions: Drug: Conventional therapy; Drug: Placebo
- intervention group: drug trimetazidine (Experimental): trimetazidine 20 mg three times Aday plus lifestyle modification
  Interventions: Drug: Trimetazidine; Drug: Conventional therapy

INTERVENTIONS:
Drug: Trimetazidine — trimetazidine at dose 20 mg three times daily to be taken by intervention group
  Arms: intervention group: drug trimetazidine
Drug: Conventional therapy — conventional therapy
Drug: Placebo — placebo tablet (inert substance has the same shape and color of intervention) to be taken by control group only
  Arms: Placebo group (conventional treatment + placebo tablet)

SUMMARY:
Objective of this study is to determine the clinical benefits of trimetazidine in improvement of MASLD

DETAILED DESCRIPTION:
the study will evaluate the possible benefits of trimetazidine when added to pateints with metabolic associated fatty liver disease

ELIGIBILITY:
Inclusion Criteria: participants were included if they met MASLD diagnostic criteria, which required imaging-confirmed hepatic steatosis (via abdominal ultrasound and CAP), along with metabolic factors (BMI ≥25 kg/m², diabetes/dysglycemia, blood pressure ≥130/85 mmHg, triglycerides ≥150 mg/dL, or reduced HDL-cholesterol)

Exclusion Criteria: The study excluded those with

* alternative steatosis causes (alcohol intake >50 g/day women or >60 g/day men
* drug-induced injury, hepatitis C, Wilson disease).
* Additional exclusion criteria covered ages below 18 years, pregnancy. decompensated cirrhosis, portal hypertension, hepatocellular carcinomas.
* Trimetazidine contraindications (Parkinson's disease, parkinsonian symptoms, tremors, severe renal impairment), patients on statins, sodium glucose transporter 2 inhibitors (SGLT2), glucagon-like peptide 1(GLP1) were among the other exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Highly sensitive CRP | measured at baseline and at six months
  Highly sensitive CRP in mg\dl by chemiillusence.
liver Fibrosis and steatosis in db./m | measured at baseline and at six months
  liver Fibrosis and steatosis in db./m fibro scan and fibro cap apparatus
ALT and AST | measured at baseline and at six months
  ALT, AST in IU/L by blood test.
Controlled attenuation parameter (CAP) | measured at baseline and at six months
  A measure of hepatic fat accumulation using transient elastography (Fibro Scan); values typically range from 100 to 400 dB/m, lower values indicate improvement Unit of measure: dB/m.
FAST Score | at baseline and at six months
  Fibro Scan-AST score; anon-invasive score to assess the risk of progressive MASH (Metabolic dysfunction-associated steatohepatitis). lower scores indicate improvement Unit of measure: Unitless index (range 0-1)

SECONDARY OUTCOMES:
LDL cholesterol | measured at baseline and at six months
  Decrease in LDL in mg\dl,
Triglyceride and total cholesterol | measured at baseline and at six months
  Triglyceride and total cholesterol in mg\dl
HOMA-IR | measured at baseline and at six months
  HOMA-IR
IL6 and TNF alpha | measured at baseline and at six months
  IL6 and TNF alpha in pg./ml by Eliza

CONTACTS AND LOCATIONS:
Overall Officials: Hoda m rabea, Assistant Professor, Principal Investigator — Beni-suaf university
Locations (1):
- Beni-Suef university, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No